CLINICAL TRIAL: NCT00396877
Title: International Randomized Double Blind Study Evaluating the Efficacy and the Safety of Clopidogrel 0.2 mg/kg Once Daily Versus Placebo in Neonates and Infants With Cyanotic Congenital Heart Disease Palliated With Systemic to Pulmonary Artery Shunt
Brief Title: Efficacy And Safety Of Clopidogrel In Neonates /Infants With Systemic To Pulmonary Artery Shunt Palliation
Acronym: CLARINET
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC5314; 2006-000946-38 (EudraCT Number)
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Heart Defects, Congenital
Keywords: cyanotic congenital heart disease; shunt palliation; thrombosis; clopidogrel
MeSH Terms: conditions — Heart Defects, Congenital; Thrombosis | interventions — Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Clopidogrel 0.2 mg/kg/day (Experimental)
  Interventions: Drug: Clopidogrel (SR25990)

INTERVENTIONS:
Drug: Clopidogrel (SR25990) — Form: reconstituted solution using Clopidogrel powder
  Route: oral or enteric
  Frequency: once daily
  Dose: daily dose adjusted for weight
  Other Names: Plavix
  Arms: Clopidogrel 0.2 mg/kg/day
Drug: placebo — Form: reconstituted solution using matching placebo powder
  Route: oral or enteric
  Frequency: once daily
  Dose: daily dose adjusted for weight
  Arms: Placebo

SUMMARY:
Contemporary management of cyanotic congenital heart disease includes three stages of surgery. Incidence of shunt thrombosis and death between the two first stages of palliation remains important.

The primary objective of the study is to evaluate the efficacy of Clopidogrel 0.2 mg/kg/day for the reduction of all cause mortality and shunt related morbidity in neonates or infants with cyanotic congenital heart disease palliated with a systemic-to-pulmonary artery shunt (e.g. modified Blalock Taussig Shunt [BTS]).

The secondary objective was to assess the safety of Clopidogrel in the study population.

DETAILED DESCRIPTION:
In this event-driven study, participants were to be randomized and treated as soon as possible after shunt placement. They were then to be treated and followed until the primary endpoint criteria was reached i.e. (shunt thrombosis, the next surgical procedure for correction of the congenital heart disease or death) or one year of age or the common study-end-date, which ever came first.

The common study-en-date was defined as the date when it was projected that 172 participants would have reached the primary endpoint criteria.

ELIGIBILITY:
Inclusion Criteria:

* Cyanotic congenital heart disease treated by any palliative systemic-to-pulmonary artery shunt.

Exclusion Criteria:

* Active bleeding or increase risk of bleeding,
* Allergy to 2 or more classes of drug,
* Unable to receive drug orally or enterically,
* Current clinically significant or persistent thrombocytopenia, neutropenia, severe hepatic or renal failure.

Max Age: 92 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 906 (Actual)
Dates: Start 2006-11; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: International Clinical Development Clinical Study Director, Study Director — Sanofi
Locations (31):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Shangaï, China
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Causeway Bay, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administraive Office, Bangkok, Thailand
- Sanofi-Aventis Admnistrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Derived] Wessel DL, Berger F, Li JS, Dahnert I, Rakhit A, Fontecave S, Newburger JW; CLARINET Investigators. Clopidogrel in infants with systemic-to-pulmonary-artery shunts. N Engl J Med. 2013 Jun 20;368(25):2377-84. doi: 10.1056/NEJMoa1114588. PMID 23782178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was initially planned with a minimum of 490 participants anticipating that it would continue until a total of 172 participants reaching primary endpoint criteria is achieved. Finally 906 participants were enrolled and randomized between November 2006 and October 2009 in 134 sites in 31 countries. Actual median follow-up was 5.8 months.
Pre-assignment Details: A participant was considered randomized when informed consent had been obtained and there was confirmation of successful allocation of a randomization number through the study treatment allocation system (Interactive Voice Response System).
Groups:
- Placebo: Reconstituted solution using Clopidogrel matching placebo powder administered once daily with a graduated syringe in the mouth or via a feeding tube.
- Clopidogrel 0.2 mg/kg/Day: Reconstituted solution using Clopidogrel powder administered once daily with a graduated syringe in the mouth or via a feeding tube.
  Route: oral or enteric
  Frequency: once daily
  Dose: daily dose adjusted for weight
Period: Overall Study
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Started | 439 (Randomized) | 467 (Randomized)
Treated | 436 | 464
Completed Treatment | 356 | 352
Completed | 433 (Completed follow-up) | 459 (Completed follow-up)
Not Completed | 6 | 8
Not completed — Lost to Follow-up | 2 | 1
Not completed — Parent(s)/guardian(s)'s request | 4 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day | Total
Number analyzed (Participants) | 439 | 467 | 906
Age, Continuous [Mean (Standard Deviation); unit: days] | 36.0 (22.5) | 36.1 (22.3) | 36.1 (22.4)
Age, Customized [Number; unit: participants]
  ≤ 30 days | 223 | 238 | 461
  30 (<) - 92 days | 216 | 229 | 445
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 198 | 383
  Male | 254 | 269 | 523
Region of Enrollment [Number; unit: participants]
  United States | 90 | 88 | 178
  Portugal | 10 | 10 | 20
  Taiwan | 12 | 10 | 22
  Hong Kong | 1 | 0 | 1
  Thailand | 2 | 3 | 5
  Spain | 16 | 14 | 30
  Israel | 3 | 4 | 7
  Russian Federation | 13 | 15 | 28
  Italy | 20 | 19 | 39
  India | 20 | 27 | 47
  France | 11 | 10 | 21
  Malaysia | 5 | 4 | 9
  Denmark | 3 | 3 | 6
  South Africa | 13 | 13 | 26
  Netherlands | 2 | 4 | 6
  China | 10 | 11 | 21
  Korea, Republic of | 3 | 2 | 5
  Finland | 2 | 1 | 3
  United Kingdom | 16 | 16 | 32
  Egypt | 4 | 6 | 10
  Hungary | 9 | 9 | 18
  Mexico | 32 | 37 | 69
  Canada | 5 | 6 | 11
  Argentina | 24 | 28 | 52
  Brazil | 31 | 34 | 65
  Belgium | 9 | 12 | 21
  Poland | 3 | 7 | 10
  Singapore | 2 | 2 | 4
  Germany | 54 | 59 | 113
  Norway | 8 | 8 | 16
  Sweden | 6 | 5 | 11
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 3.5 (0.7) | 3.4 (0.7) | 3.5 (0.7)
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 51.8 (4.6) | 51.4 (4.4) | 51.6 (4.5)
Type of systemic-to-pulmonary artery shunt palliation [Number; unit: participants] — One participant didn't have a systemic-to-pulmonary artery shunt but underwent stenting of the right ventricular outflow track.
  participants
    Modified Blalock Taussig Shunt with Norwood | 51 | 62 | 113
    Modified Blalock Taussig Shunt without Norwood | 252 | 257 | 509
    Sano procedure with Norwood | 54 | 60 | 114
    Sano procedure without Norwood | 2 | 5 | 7
    Central shunt | 38 | 40 | 78
    Stent of ductus arteriosus | 42 | 42 | 84
    Not applicable | 0 | 1 | 1
Shunt on cardiopulmonary bypass [Number; unit: participants]
  Yes | 177 | 194 | 371
  No | 262 | 273 | 535
Age at shunt palliation [Mean (Standard Deviation); unit: days] | 16.0 (18.7) | 16.2 (18.6) | 16.1 (18.7)
Time from shunt palliation to randomization [Number; unit: participants]
  ≤ 1 week | 116 | 113 | 229
  1 (<) to 2 weeks | 105 | 126 | 231
  2 (<) to 4 weeks | 117 | 119 | 236
  > 4 weeks | 101 | 109 | 210

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reaching Primary Endpoint Criteria (First Occurrence of Death / Shunt Thrombosis / Cardiac Procedure < 120 Days Considered of Thrombotic Nature)
Description: The primary endpoint was the first occurence of any of the following events: Death (including heart transplant); Shunt thrombosis requiring intervention; Hospitalization for bi-directional Glenn procedure or any cardiac related intervention prior to 120 days of age following an event or a shunt narrowing considered to be of thrombotic nature by the blinded adjudication committee.
  Only the first event was counted.
Time Frame: Median follow-up of 5.8 months (up to a maximum of 12 months after randomization)
Population: The analysis was performed on the intent-to-treat (ITT) population (i.e. all randomized participants irrespective of whether or not the participant actually received study drug or the participant's compliance with the study protocol). Participants were included in the treatment group to which they were originally allocated.
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 439 | 467
participants
  Death / Shunt Thrombosis / Cardiac Procedure | 90 | 89
  - Death | 60 | 51
  - Shunt thrombosis | 21 | 26
  - Cardiac procedure <120 days of thrombotic nature | 9 | 12
Statistical Analysis 1: Comparison: Placebo vs Clopidogrel 0.2 mg/kg/Day; Due to the limited knowledge in this population, 3 interim analyses were performed at approximatively 40%, 60%, 80% and 100% of of the maximum number of 172 required primary efficacy events to evaluate the effect of Clopidogrel on the primary endpoint with the potential to end the trial in case of a clear efficacy advantage for Clopidogrel. The study was designed with 80% power and an overall type I error rate of 5%; Test type: Superiority or Other; p = 0.4340, Log Rank — The a-priori threshold for statistical significance was < 0.035 reflecting the adjustment for interim analyses. No other adjustment for multiplicity was made; A two-sided log-rank test was used; Relative Risk Reduction (%) = 11.1, 95% CI 2-sided [-19.2 to 33.6] — The Relative Risk Reduction (Clopidogrel versus placebo) and its corresponding 95% confidence interval were estimated using Cox's proportional hazards model

2. Secondary Outcome: Number of Participants With Bleeding Events
Description: Bleeding events spanning from signature of the Informed Consent Form up to the last visit were collected as for any Adverse Event.
  The 'on-treatment' period was defined as the period from randomization up until 28 days after treatment discontinuation or final follow-up visit, whichever came first, and participants who experienced bleeding events during that period were counted.
Time Frame: From randomization up to 28 days after treatment discontinuation or final follow-up visit, whichever comes first
Population: The analysis was performed on the exposed population (i.e. all randomized participants who received at least one dose of study drug regardless of the amount of treatment received). Participants were included in the treatment group according to the treatment received.
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 436 | 464
participants
  Any bleeding event | 88 | 87
  - Serious | 32 | 30
  - Serious with an outcome of death | 1 | 1
  - Leading to permanent treatment discontinuation | 9 | 9

3. Secondary Outcome: Number of Participants According to Bleeding Type/Etiology
Description: For all reported bleeding events, the type and the etiology of the bleeding event were collected. Participants who experienced bleeding events during the 'on-treatment period' were counted by bleeding type and etiology. Participants who had multiple bleedings could be counted several times.
Time Frame: From randomization up to 28 days after treatment discontinuation or final follow-up visit, whichever comes first
Population: The analysis was performed on the same population as previously (i.e. exposed population).
Measure: Number; unit: participants
Arm/Group | Placebo | Clopidogrel 0.2 mg/kg/Day
Number analyzed (Participants) | 436 | 464
participants
  Spontaneous | 60 | 56
  Post-traumatic | 6 | 11
  Puncture (vascular access site) | 19 | 9
  Surgical | 10 | 17

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent Form up to the last visit were collected.
Description: The analysis was performed on the exposed population and included all AE that developed/worsened during the 'on-treatment period' (i.e. from randomization up to 28 days after treatment discontinuation or final follow-up visit, whichever came first).
Arm/Group | Placebo | Clopidogrel 0.2mg/kg/Day
Serious Adverse Events (participants affected / at risk) | 196/436 | 234/464
Other Adverse Events (participants affected / at risk) | 96/436 | 107/464
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=436) | Clopidogrel 0.2mg/kg/Day (N=464)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 13 | 11
GASTROENTERITIS (Infections and infestations) | 14 | 24
PNEUMONIA (Infections and infestations) | 9 | 21
BRONCHIOLITIS (Infections and infestations) | 12 | 15
URINARY TRACT INFECTION (Infections and infestations) | 6 | 6
VIRAL INFECTION (Infections and infestations) | 6 | 7
BRONCHITIS (Infections and infestations) | 1 | 4
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 3
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 2 | 7
WOUND INFECTION (Infections and infestations) | 2 | 3
INFLUENZA (Infections and infestations) | 5 | 6
GASTROENTERITIS VIRAL (Infections and infestations) | 4 | 5
RESPIRATORY TRACT INFECTION (Infections and infestations) | 3 | 3
SEPSIS (Infections and infestations) | 4 | 8
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 1
EAR INFECTION (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 4 | 4
OTITIS MEDIA (Infections and infestations) | 1 | 1
PULMONARY SEPSIS (Infections and infestations) | 3 | 5
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 3
ENDOCARDITIS (Infections and infestations) | 1 | 4
LOWER RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 2
RESPIRATORY SYNCYTIAL VIRUS INFECTION (Infections and infestations) | 3 | 4
SKIN INFECTION (Infections and infestations) | 0 | 2
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 | 4
LUNG INFECTION (Infections and infestations) | 2 | 3
NOSOCOMIAL INFECTION (Infections and infestations) | 0 | 2
RESPIRATORY SYNCYTIAL VIRUS BRONCHIOLITIS (Infections and infestations) | 1 | 2
RHINITIS (Infections and infestations) | 0 | 1
BRONCHITIS BACTERIAL (Infections and infestations) | 0 | 1
BRONCHITIS VIRAL (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1 | 2
ENTEROCOCCAL BACTERAEMIA (Infections and infestations) | 2 | 2
FUNGAL SEPSIS (Infections and infestations) | 0 | 2
GASTROENTERITIS ADENOVIRUS (Infections and infestations) | 1 | 1
GASTROENTERITIS ROTAVIRUS (Infections and infestations) | 3 | 2
LARYNGITIS (Infections and infestations) | 0 | 1
PNEUMONIA RESPIRATORY SYNCYTIAL VIRAL (Infections and infestations) | 0 | 2
POST PROCEDURAL INFECTION (Infections and infestations) | 1 | 2
PYELONEPHRITIS (Infections and infestations) | 2 | 2
ROTAVIRUS INFECTION (Infections and infestations) | 1 | 1
SEPTIC SHOCK (Infections and infestations) | 0 | 2
UROSEPSIS (Infections and infestations) | 1 | 2
VIRAL RASH (Infections and infestations) | 0 | 2
ABDOMINAL SEPSIS (Infections and infestations) | 0 | 1
BACTERIAL INFECTION (Infections and infestations) | 0 | 1
BACTERIAL SEPSIS (Infections and infestations) | 2 | 0
CATHETER SEPSIS (Infections and infestations) | 4 | 1
CELLULITIS (Infections and infestations) | 0 | 1
ENTEROBACTER SEPSIS (Infections and infestations) | 1 | 1
ENTEROCOCCAL INFECTION (Infections and infestations) | 1 | 0
ESCHERICHIA SEPSIS (Infections and infestations) | 0 | 1
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
HAEMOPHILUS INFECTION (Infections and infestations) | 0 | 1
IMPETIGO (Infections and infestations) | 0 | 1
INCISION SITE INFECTION (Infections and infestations) | 2 | 1
KLEBSIELLA BACTERAEMIA (Infections and infestations) | 0 | 1
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0
MEDIASTINAL ABSCESS (Infections and infestations) | 0 | 1
MENINGITIS PNEUMOCOCCAL (Infections and infestations) | 1 | 1
PARAINFLUENZAE VIRUS INFECTION (Infections and infestations) | 1 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 0 | 1
PNEUMONIA ESCHERICHIA (Infections and infestations) | 0 | 1
PNEUMONIA VIRAL (Infections and infestations) | 0 | 1
PSEUDOMONAL SEPSIS (Infections and infestations) | 1 | 0
SEPSIS SYNDROME (Infections and infestations) | 0 | 1
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ADENOVIRUS INFECTION (Infections and infestations) | 1 | 0
CANDIDA SEPSIS (Infections and infestations) | 1 | 0
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1 | 0
GASTROENTERITIS CALICIVIRAL (Infections and infestations) | 1 | 0
GASTROINTESTINAL INFECTION (Infections and infestations) | 1 | 0
KLEBSIELLA SEPSIS (Infections and infestations) | 1 | 0
LOCALISED INFECTION (Infections and infestations) | 1 | 0
MEDIASTINITIS (Infections and infestations) | 3 | 0
MENINGITIS ASEPTIC (Infections and infestations) | 1 | 0
OTITIS MEDIA ACUTE (Infections and infestations) | 2 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 1 | 0
PNEUMONIA INFLUENZAL (Infections and infestations) | 1 | 0
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 2 | 0
POST PROCEDURAL CELLULITIS (Infections and infestations) | 1 | 0
PYELONEPHRITIS ACUTE (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 | 0
VIRAL DIARRHOEA (Infections and infestations) | 1 | 0
WOUND ABSCESS (Infections and infestations) | 2 | 0
WOUND SEPSIS (Infections and infestations) | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 3 | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 2
DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
DISSEMINATED INTRAVASCULAR COAGULATION (Blood and lymphatic system disorders) | 1 | 0
HAEMORRHAGIC ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
MILK ALLERGY (Immune system disorders) | 0 | 1
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 1 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 6
FEEDING DISORDER OF INFANCY OR EARLY CHILDHOOD (Metabolism and nutrition disorders) | 5 | 2
WEIGHT GAIN POOR (Metabolism and nutrition disorders) | 3 | 0
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 6 | 3
FOOD INTOLERANCE (Metabolism and nutrition disorders) | 3 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 | 1
MALNUTRITION (Metabolism and nutrition disorders) | 0 | 1
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 2 | 2
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOGLYCAEMIC SEIZURE (Metabolism and nutrition disorders) | 1 | 0
AGITATION (Psychiatric disorders) | 1 | 1
CONVULSION (Nervous system disorders) | 2 | 3
PARTIAL SEIZURES (Nervous system disorders) | 0 | 3
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 3
VOCAL CORD PARALYSIS (Nervous system disorders) | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 2
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 | 2
LETHARGY (Nervous system disorders) | 0 | 2
POOR SUCKING REFLEX (Nervous system disorders) | 0 | 1
VOCAL CORD PARESIS (Nervous system disorders) | 0 | 1
CLONIC CONVULSION (Nervous system disorders) | 0 | 1
DYSKINESIA (Nervous system disorders) | 0 | 1
EMBOLIC STROKE (Nervous system disorders) | 0 | 1
ENCEPHALITIS (Nervous system disorders) | 0 | 1
HYPOGLYCAEMIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 1
ISCHAEMIC CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1
PHRENIC NERVE PARALYSIS (Nervous system disorders) | 0 | 1
SUBARACHNOID HAEMORRHAGE NEONATAL (Nervous system disorders) | 0 | 1
CONVULSIONS LOCAL (Nervous system disorders) | 1 | 0
FEBRILE CONVULSION (Nervous system disorders) | 1 | 0
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
MIDDLE EAR INFLAMMATION (Ear and labyrinth disorders) | 0 | 1
CYANOSIS (Cardiac disorders) | 9 | 24
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 4
CARDIAC FAILURE (Cardiac disorders) | 5 | 6
BRADYCARDIA (Cardiac disorders) | 4 | 3
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 4
CARDIAC ARREST (Cardiac disorders) | 2 | 3
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1 | 4
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 3
RIGHT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 2
ARRHYTHMIA (Cardiac disorders) | 0 | 2
ATRIOVENTRICULAR BLOCK (Cardiac disorders) | 0 | 2
CARDIAC PERFORATION (Cardiac disorders) | 0 | 1
ATRIOVENTRICULAR BLOCK COMPLETE (Cardiac disorders) | 1 | 0
CARDIAC DISORDER (Cardiac disorders) | 0 | 1
CARDIAC FAILURE ACUTE (Cardiac disorders) | 0 | 1
CARDIAC PSEUDOANEURYSM (Cardiac disorders) | 0 | 1
CARDIOGENIC SHOCK (Cardiac disorders) | 2 | 1
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 | 1
DILATATION VENTRICULAR (Cardiac disorders) | 0 | 1
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 | 1
PERICARDIAL HAEMORRHAGE (Cardiac disorders) | 1 | 1
PULMONARY VALVE STENOSIS (Cardiac disorders) | 3 | 1
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 0 | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 | 1
LOW CARDIAC OUTPUT SYNDROME (Cardiac disorders) | 2 | 0
NODAL ARRHYTHMIA (Cardiac disorders) | 1 | 0
TRICUSPID VALVE INCOMPETENCE (Cardiac disorders) | 3 | 0
VENTRICULAR DYSFUNCTION (Cardiac disorders) | 1 | 0
AORTIC STENOSIS (Vascular disorders) | 2 | 2
VENA CAVA THROMBOSIS (Vascular disorders) | 1 | 2
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 0 | 1
SHOCK (Vascular disorders) | 0 | 1
VASCULAR STENOSIS (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 1 | 0
EMBOLISM (Vascular disorders) | 1 | 0
HYPOTENSION (Vascular disorders) | 2 | 0
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 1 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 11 | 14
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 3 | 5
PULMONARY ARTERY STENOSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 3
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 4 | 5
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 2 | 3
DIAPHRAGMATIC PARALYSIS (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 2 | 2
STRIDOR (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 2
LARYNGEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OBSTRUCTIVE AIRWAYS DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 2 | 2
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY VEIN STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
TACHYPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ACUTE RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 2 | 1
BRONCHOSTENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CHYLOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY VEIN OCCLUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 1 | 1
RESPIRATORY FATIGUE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
TRACHEOMALACIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL HAEMATOMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
MEDIASTINAL HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 | 0
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOCAL CORD THICKENING (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VOMITING (Gastrointestinal disorders) | 5 | 5
DIARRHOEA (Gastrointestinal disorders) | 1 | 5
HAEMATOCHEZIA (Gastrointestinal disorders) | 7 | 2
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 4 | 6
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 2 | 4
NECROTISING COLITIS (Gastrointestinal disorders) | 1 | 6
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 2
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 1
DYSPHAGIA (Gastrointestinal disorders) | 2 | 3
ENTEROCOLITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 2
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 1
ANAL FISSURE (Gastrointestinal disorders) | 1 | 0
ENTEROCOLITIS (Gastrointestinal disorders) | 1 | 0
GASTRITIS (Gastrointestinal disorders) | 0 | 1
HAEMATEMESIS (Gastrointestinal disorders) | 1 | 1
LOWER GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 3 | 1
POST-TUSSIVE VOMITING (Gastrointestinal disorders) | 0 | 1
DUODENAL STENOSIS (Gastrointestinal disorders) | 1 | 0
ENTERITIS (Gastrointestinal disorders) | 2 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 1 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
INTESTINAL PERFORATION (Gastrointestinal disorders) | 1 | 0
PNEUMATOSIS INTESTINALIS (Gastrointestinal disorders) | 1 | 0
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 | 0
ACUTE HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 1
DERMATITIS DIAPER (Skin and subcutaneous tissue disorders) | 0 | 1
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 | 1
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 1
SUBCUTANEOUS EMPHYSEMA (Skin and subcutaneous tissue disorders) | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 2
HAEMATURIA (Renal and urinary disorders) | 0 | 1
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 1 | 0
BLADDER PROLAPSE (Renal and urinary disorders) | 1 | 0
VESICOURETERIC REFLUX (Renal and urinary disorders) | 1 | 0
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 | 2
COARCTATION OF THE AORTA (Congenital, familial and genetic disorders) | 2 | 1
LARYNGOMALACIA (Congenital, familial and genetic disorders) | 0 | 1
PULMONARY ARTERY STENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 0 | 1
PYLORIC STENOSIS (Congenital, familial and genetic disorders) | 1 | 1
PYREXIA (General disorders) | 3 | 5
PUNCTURE SITE HAEMORRHAGE (General disorders) | 2 | 1
CATHETER RELATED COMPLICATION (General disorders) | 1 | 1
CATHETER SITE HAEMORRHAGE (General disorders) | 0 | 1
IRRITABILITY (General disorders) | 0 | 1
CATHETER THROMBOSIS (General disorders) | 1 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
FEELING ABNORMAL (General disorders) | 1 | 0
VESSEL PUNCTURE SITE HAEMATOMA (General disorders) | 1 | 0
OXYGEN SATURATION DECREASED (Investigations) | 10 | 11
BLOOD URINE PRESENT (Investigations) | 1 | 0
PULMONARY ARTERIAL PRESSURE DECREASED (Investigations) | 0 | 1
WEIGHT INCREASED (Investigations) | 0 | 1
ASPIRATION BRONCHIAL (Investigations) | 1 | 0
OXYGEN SATURATION INCREASED (Investigations) | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 1 | 0
PULMONARY ARTERIAL PRESSURE INCREASED (Investigations) | 1 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 4 | 8
ACCIDENTAL OVERDOSE (Injury, poisoning and procedural complications) | 2 | 3
OPERATIVE HAEMORRHAGE (Injury, poisoning and procedural complications) | 3 | 3
POSTOPERATIVE FEVER (Injury, poisoning and procedural complications) | 0 | 1
SHUNT STENOSIS (Injury, poisoning and procedural complications) | 2 | 2
FALL (Injury, poisoning and procedural complications) | 0 | 1
SUTURE RELATED COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
FEEDING TUBE COMPLICATION (Injury, poisoning and procedural complications) | 0 | 1
PNEUMOTHORAX TRAUMATIC (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 1
POST VACCINATION SYNDROME (Injury, poisoning and procedural complications) | 0 | 1
PROCEDURAL SITE REACTION (Injury, poisoning and procedural complications) | 1 | 1
SHUNT BLOOD FLOW EXCESSIVE (Injury, poisoning and procedural complications) | 0 | 1
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 | 0
DEVICE BREAKAGE (Injury, poisoning and procedural complications) | 1 | 0
DRUG TOXICITY (Injury, poisoning and procedural complications) | 1 | 0
GRAFT THROMBOSIS (Injury, poisoning and procedural complications) | 1 | 0
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE RESPIRATORY DISTRESS (Injury, poisoning and procedural complications) | 1 | 0
POSTOPERATIVE WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 2 | 0
SEROMA (Injury, poisoning and procedural complications) | 1 | 0
SHUNT MALFUNCTION (Injury, poisoning and procedural complications) | 3 | 0
SHUNT OCCLUSION (Injury, poisoning and procedural complications) | 1 | 0
SKULL FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
SUTURE RUPTURE (Injury, poisoning and procedural complications) | 1 | 0
VASCULAR PSEUDOANEURYSM (Injury, poisoning and procedural complications) | 1 | 0
ANORECTAL OPERATION (Surgical and medical procedures) | 0 | 1
CARDIOVASCULAR EVENT PROPHYLAXIS (Surgical and medical procedures) | 0 | 1
URETERONEOCYSTOSTOMY (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=436) | Clopidogrel 0.2mg/kg/Day (N=464)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 | 60
NASOPHARYNGITIS (Infections and infestations) | 24 | 21
VOMITING (Gastrointestinal disorders) | 18 | 32
DIARRHOEA (Gastrointestinal disorders) | 20 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the Investigator can publish the results. Prior to publication, the sponsor shall review the manuscript and can request changes, provided they do not jeopardize the accuracy and/or the scientific value of the publication. The approval is given in writing by the sponsor, not exceeding 90 days.